CLINICAL TRIAL: NCT02823600
Title: A Feasibility Study of Retinal Screening Using the RetinaVue 100 Hand- Held (Non-mydriatic) Camera in Outpatient Dialysis Centers
Brief Title: Feasibility Study of Retinal Screening Using the RetinaVue 100 Camera in Outpatient Dialysis Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Welch Allyn (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 16-1116
Record Dates: First submitted 2016-06-30; First posted 2016-07-06 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-06

CONDITIONS: Kidney Failure, Chronic; Eye Diseases; Diabetic Retinopathy
Keywords: retinal screening; outpatient dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Eye Diseases; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RetinaVue 100 camera (Other): Participants will have a retinal screening completed by study staff using the FDA-approved RetinaVue 100 hand-held camera
  Interventions: Device: RetinaVue 100 camera

INTERVENTIONS:
Device: RetinaVue 100 camera — Images of the subject's eye will be obtained using the RetinaVue 100 camera and uploaded to a secure network. The study doctor, a board-certified ophthalmologist, will interpret the patient images and return a diagnosis and management plan to the dialysis unit.

SUMMARY:
The purpose of this research study is to look at retinal abnormalities in outpatient renal dialysis patients using the FDA approved RetinaVue 100 hand-held (non-mydriatic) camera.

DETAILED DESCRIPTION:
There are no studies evaluating (diabetic or non-diabetic) retinopathy in the renal dialysis patient population (~300,000 Americans). Approximately 50% of this population has End-stage Retinal Disease (ESRD) due to diabetes. Dialysis patients are among the most debilitated patients, and thus, have even more barriers to receiving their recommended annual retinal evaluation. The advent of the RetinaVue hand-held retinal camera holds great promise in this population, as dialysis patients access medical care 3 times a week, for several hours at a time at their dialysis clinic.

ELIGIBILITY:
Inclusion Criteria:

* The subject must currently be seeking treatment for end-stage renal disease (ESRD) at one of the specified dialysis clinics.
* The subject must be ≥ 18 years of age.

Exclusion Criteria:

* The subject is <18 years of age.
* No exclusions will be made on the basis of gender, ethnicity, or race.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Garg, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Ophthalmology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- RetinaVue 100 Camera: Participants will have a retinal exam completed by study staff using the FDA-approved RetinaVue 100 hand-held camera
  RetinaVue 100 camera: Images of the subject's retina will be obtained using the RetinaVue 100 camera and uploaded to a secure network. The study doctor, a board-certified ophthalmologist, will interpret the patient images and return a diagnosis and management plan to the dialysis unit.
Period: Overall Study
Arm/Group | RetinaVue 100 Camera
Started | 68
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- RetinaVue 100 Camera: All participants will have a retinal eye exam completed by study staff using the FDA-approved RetinaVue 100 hand-held camera
Arm/Group | RetinaVue 100 Camera
Number analyzed (Participants) | 68
Age, Customized [Mean (Standard Deviation); unit: years] — This measure is divided into categories by referral status, which is used as a proxy for retinal disease severity. With "no retinopathy" as the least severe or no disease and "retinopathy with referral" as the most severe.
  years
    No retinopathy | 54.7 (18.1)
    Retinopathy without referral | 60.0 (6.6)
    Retinopathy with referral | 57.1 (11.6)
Sex/Gender, Customized [Count of Participants; unit: Participants] — This measure is divided into categories by referral status, which is used as a proxy for retinal disease severity. With "no retinopathy" as the least severe or no disease and "retinopathy with referral" as the most severe.
  Participants
    Female : No retinopathy | 17
    Female : Retinopathy without referral | 6
    Female : Retinopathy with referral | 6
    Male : No retinopathy | 16
    Male : Retinopathy without referral | 5
    Male : Retinopathy with referral | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — This measure is divided into categories by referral status, which is used as a proxy for retinal disease severity. With "no retinopathy" as the least severe or no disease and "retinopathy with referral" as the most severe.
  Participants
    African American: No retinopathy | 14
    African American: Retinopathy without referral | 6
    African American: Retinopathy with referral | 11
    Caucasian: No retinopathy | 11
    Caucasian: Retinopathy without referral | 3
    Caucasian: Retinopathy with referral | 8
    Hispanic: No retinopathy | 8
    Hispanic: Retinopathy without referral | 2
    Hispanic: Retinopathy with referral | 4
    Data Missing | 1
End-Stage Renal Disease Etiology [Count of Participants; unit: Participants] — This measure is divided into categories by referral status, which is used as a proxy for retinal disease severity. With "no retinopathy" as the least severe or no disease and "retinopathy with referral" as the most severe.
  Participants
    Diabetes: No retinopathy | 7
    Diabetes: Retinopathy without referral | 8
    Diabetes: Retinopathy with referral | 13
    Hypertension: No retinopathy | 12
    Hypertension: Retinopathy without referral | 1
    Hypertension: Retinopathy with referral | 7
    Other: No retinopathy | 13
    Other: Retinopathy without referral | 2
    Other: Retinopathy with referral | 4
    Data Missing | 7
Diabetic dialysis population [Count of Participants; unit: Participants] — Proportion of entire study population with a diabetes mellitus (DM) diagnosis.
  Participants
    Diabetes: Yes | 37
    Diabetes: No | 31

OUTCOME MEASURES:

1. Primary Outcome: Usability of the RetinaVue Hand-Held 100 Camera
Description: Usability of RetinaVue camera assessed by determining the number and percentage of inadequate images and the number and percentage of adequate images.
Time Frame: baseline visit
Measure: Count of Units; unit: Retinal Images
Units Other Than Participants: Retinal Images
Groups:
- Images: This group is the total number of images, 136, captured from the study population.
Arm/Group | Images
Number analyzed (Participants) | 68
Number analyzed (Retinal Images) | 136
Retinal Images
  Inadequate Images | 20
  Adequate Images | 116

2. Secondary Outcome: Overall Retinopathy in a Dialysis Population
Description: Number of participants found to have retinopathy in a dialysis population
Time Frame: Post retinal eye exam
Measure: Count of Participants; unit: Participants
Groups:
- RetinaVue 100 Camera: All participants will have a retinal exam completed by study staff using the FDA-approved RetinaVue 100 hand-held camera
Arm/Group | RetinaVue 100 Camera
Number analyzed (Participants) | 68
Participants
  No retinopathy | 33
  Retinopathy | 35

3. Secondary Outcome: Participant Satisfaction
Description: Participant satisfaction survey data to be collected following the completion of retinal eye exam. Participants will be assessed on participant satisfaction measures such as comfort of experience, recovery time, and time invested in undergoing procedure vs. traditional retinal exam methods. The survey utilized a five-point Likert scale with the following responses: (1) strongly agree, (2) agree, (3) neutral, (4) disagree, (5) strongly disagree. The outcome measure is reported percentages for each of the six survey components.
Time Frame: Post retinal eye exam
Population: This analysis is based on responses from the 39 that completed the survey.
Measure: Number; unit: Percentage of participants
Arm/Group | RetinaVue 100 Camera
Number analyzed (Participants) | 39
Percentage of participants
  Satisfied time complete eye exam:Strongly agree | 61.5
  Satisfied time complete eye exam : Agree | 28.2
  Satisfied time complete eye exam : Neutral | 10.3
  Satisfied time complete eye exam:Disagree | 0
  Satisfied time complete eye exam:Strongly Disagree | 0
  Comfort during eye exam : Strongly agree | 75.4
  Comfort during eye exam : Agree | 24.6
  Comfort during eye exam : Neutral | 0
  Comfort during eye exam : Disagree | 0
  Comfort during eye exam : Strongly Disagree | 0
  Comfort after eye exam : Strongly agree | 82.0
  Comfort after eye exam : Agree | 18.0
  Comfort after eye exam : Neutral | 0
  Comfort after eye exam : Disagree | 0
  Comfort after eye exam : Strongly Disagree | 0
  1st eye quick recovery:Strongly agree | 53.9
  1st eye quick recovery:Agree | 41.0
  1st eye quick recovery:Neutral | 5.1
  1st eye quick recovery:Disagree | 0
  1st eye quick recovery:Strongly Disagree | 0
  2nd eye quick recovery:Strongly agree | 59.0
  2nd eye quick recovery:Agree | 35.9
  2nd eye quick recovery:Neutral | 5.1
  2nd eye quick recovery :Disagree | 0
  2nd eye quick recovery:Strongly Disagree | 0
  Satisfied w overall experience:Strongly agree | 79.5
  Satisfied w overall experience:Agree | 20.5
  Satisfied w overall experience:Neutral | 0
  Satisfied w overall experience:Disagree | 0
  Satisfied w overall experience:Strongly Disagree | 0

4. Secondary Outcome: Pre-and Post-eye Exam Rates in the Diabetic Dialysis Population
Description: Changes in eye exam rates of the diabetic subset of total population from baseline (i.e. study entry) and post-enrollment in study. Baseline data were to be obtained from the UNC electronic medical record (EMR) as the number of participants with eye exams within the past year and post data would consist of the number of participants completing a study exam.
Time Frame: Baseline and post retinal eye exam
Population: Baseline retinal examination data were not present within the EMR; therefore, this analysis could not be performed.
Arm/Group | RetinaVue 100 Camera
Number analyzed (Participants) | 0

5. Post Hoc Outcome: Number of Diabetic Dialysis Subjects Undergoing Retinal Exam During Study Using the RetinaVue 100 Camera
Time Frame: Up to as much as one year after study enrollment
Population: Diabetic dialysis participants
Measure: Count of Participants; unit: Participants
Arm/Group | RetinaVue 100 Camera
Number analyzed (Participants) | 37
Participants
  No retinopathy | 11
  Retinopathy without referral | 9
  Retinopathy with referral | 17

ADVERSE EVENTS:
Time Frame: The duration of the eye exam and the period following, up to a two hour interval.
Groups:
- ESRD: This study only had only one arm. All those individuals who met eligibility criteria and provided voluntary consent, were enrolled to this study and followed the same procedures.
Arm/Group | ESRD
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 0/68

LIMITATIONS AND CAVEATS:
Limitations included small sample size which led to low power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT02823600/Prot_SAP_000.pdf